CLINICAL TRIAL: NCT02727751
Title: An Open Label Long-Term Safety Study of Tenapanor for the Treatment of Constipation-Predominant Irritable Bowel Syndrome (IBS-C)
Brief Title: A Long-Term Safety Study of Tenapanor for the Treatment of IBS-C
Acronym: T3MPO-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ardelyx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TEN-01-303
Record Dates: First submitted 2016-03-23; First posted 2016-04-05 (Estimated); Results first posted 2020-04-24 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-08

CONDITIONS: Constipation Predominant Irritable Bowel Syndrome
MeSH Terms: interventions — tenapanor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 50mg BID (Experimental): Tenapanor, 50 mg BID (100 mg total)
  Interventions: Drug: Tenapanor

INTERVENTIONS:
Drug: Tenapanor
  Other Names: RDX5791; AZD1722

SUMMARY:
This phase 3, open label study will evaluate the safety of tenapanor 50 mg BID in subjects with constipation-predominant irritable bowel syndrome (IBS-C) defined by the ROME III criteria. Subjects who have completed either TEN-01-301 (16 weeks) or TEN-01-302 (26 weeks) studies may be enrolled. Subjects will take tenapanor for approximately 52-55 weeks total based on previous protocol and this study.

DETAILED DESCRIPTION:
During the treatment period of up to 39-weeks, subjects will return for study visits approximately every 13 weeks. Subjects will undergo safety assessments at these visits, which may include a physical exam, ECG, vital signs, and clinical labs. Adverse events and concomitant medications will be recorded. Medication compliance will be monitored and the subjects will be given additional study drug as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Subjects completed all 16 weeks of TEN-01-301 or all 26 weeks of TEN-01-302
* Subject demonstrated adequate compliance with the study procedures during either the TEN-01-301 or TEN-01-302 studies
* Females must be of non-childbearing potential; If of child-bearing potential, must have negative pregnancy test and confirm the use of one of the appropriate means of contraception
* Males must agree to use appropriate methods of barrier contraception or have documented surgical sterilization

Exclusion Criteria:

* Subject has been withdrawn or discontinued prematurely from either TEN-01-301 or TEN-01-302
* The subject reports using any prohibited medication and is not willing to abide by the restrictions for intake
* Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2016-03; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David P Rosenbaum, Ph.D., Study Chair — Ardelyx, Inc.
Locations (1):
- Ardelyx Clinical Site, Miami, Florida, United States

REFERENCES:
- [Derived] Lembo AJ, Friedenberg KA, Fogel RP, Edelstein S, Zhao S, Yang Y, Rosenbaum DP, Chey WD. Long-term safety of tenapanor in patients with irritable bowel syndrome with constipation in the T3MPO-3 study. Neurogastroenterol Motil. 2023 Nov;35(11):e14658. doi: 10.1111/nmo.14658. Epub 2023 Sep 5. PMID 37668173
- [Derived] Chey WD, Lembo AJ, Yang Y, Rosenbaum DP. Efficacy of Tenapanor in Treating Patients With Irritable Bowel Syndrome With Constipation: A 26-Week, Placebo-Controlled Phase 3 Trial (T3MPO-2). Am J Gastroenterol. 2021 Jun 1;116(6):1294-1303. doi: 10.14309/ajg.0000000000001056. PMID 33337659

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 50mg BID
Started | 312
Completed | 262
Not Completed | 50

BASELINE CHARACTERISTICS:
Arm/Group | 50mg BID
Number analyzed (Participants) | 312
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (13.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 255
  Male | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 130
  Not Hispanic or Latino | 182
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 89
  White | 217
  More than one race | 2
  Unknown or Not Reported | 2
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.98 (6.707)

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events in >2% Patients
Description: Safety assessments will be based on adverse events, clinical laboratory tests, vital signs, ECG, and physical exams
Time Frame: 52-55 weeks
Measure: Number; unit: participants
Arm/Group | 50mg BID
Number analyzed (Participants) | 312
participants
  Diarrhea | 33
  Flatulence | 7
  Upper Respiratory Tract Infection | 7
  Headache | 11

ADVERSE EVENTS:
Time Frame: This was an extension study that ran for up to 1 year
Arm/Group | 50mg BID
All-Cause Mortality (participants affected / at risk) | 0/312
Serious Adverse Events (participants affected / at risk) | 3/312
Other Adverse Events (participants affected / at risk) | 33/312
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50mg BID (N=312)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50mg BID (N=312)
Diarrhea (Gastrointestinal disorders) | 33 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-01-29): https://cdn.clinicaltrials.gov/large-docs/51/NCT02727751/Prot_000.pdf
  • Statistical Analysis Plan (2016-03-08): https://cdn.clinicaltrials.gov/large-docs/51/NCT02727751/SAP_001.pdf